CLINICAL TRIAL: NCT02200341
Title: MBCT Effects on Brain Mechanisms of Interoceptive Awareness and Rumination in MDD
Brief Title: Effects of Mindfulness-based Cognitive Therapy on Brain Mechanisms in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Desbordes, Gaelle, Instructor in Radiology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014P000223; K01AT008225 (NIH)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): Mindfulness-Based Cognitive Therapy (MBCT) 8-week intervention
  Interventions: Behavioral: MBCT
- Progressive Relaxation Training - Psychoeducation (Active Comparator): Progressive Relaxation Training and Psychoeducation (PRT-PsyEd) 8-week intervention
  Interventions: Behavioral: PRT-PsyEd

INTERVENTIONS:
Behavioral: MBCT
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: PRT-PsyEd
  Arms: Progressive Relaxation Training - Psychoeducation

SUMMARY:
The purpose of this study is to investigate the effects of Mindfulness-Based Cognitive Therapy (MBCT) on brain mechanisms associated with interoceptive awareness and rumination in individuals suffering from major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* current mild-to-moderate depression symptoms (score 12-36 on IDS-C30)
* history of at least 3 depressive episodes or history of 2 years of depression symptoms
* on either no pharmacological treatment or on maintenance antidepressant treatment for at least 8 weeks before the start of the intervention
* English literacy
* normal or near-normal vision

Exclusion Criteria:

i. A score of 37 of higher on the Inventory of Depressive Symptomatology - Clinician version (IDS-C30).

ii. Significant risk for suicide, defined by a score of 3 on Item 18 in the IDS-C30, or as assessed by evaluating clinician.

iii. Severe and unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.

iv. The following DSM disorders: any bipolar disorder (current or past), a primary psychotic disorder (current or past), or current psychotic symptoms. However, entry of patients with anxiety disorder(s) will be permitted if the depressive disorder is judged to be the predominant disorder.

v. Active diagnosis of substance abuse or dependence disorders within the last 3 months.

vi. General conditions that would impede participation in a group intervention, as assessed by the evaluating clinician or the therapist delivering the MBCT intervention (such as severe characterological disorders, cognitive impairment, tendencies toward physical aggression).

vii. Past or current training in mindfulness (MBCT, Mindfulness-Based Stress Reduction) or in the Relaxation Response.

viii. Significant training in meditation (or related practices), i.e., more than 10 meditation classes in the past 3 months, or more than 10 classes in yoga, Tai Chi, or Qi Gong in the past 3 months.

ix. Currently taking any psychoactive drugs (whether prescription, over-the-counter, or recreational) other than prescribed antidepressants. This restriction includes the following supplements: Hypericum perforatum (St. John's wort), Valeriana officinalis (valerian), and 5-Hydroxytryptophan (5-HTP).

x. Any change in type or dosage of treatment (whether with antidepressant medication or with psychotherapy or psychosocial intervention) in the 8 weeks preceding the start of the intervention.

xi. Standard exclusion criteria for undergoing magnetic resonance imaging (MRI) procedures for research purposes, i.e., Meniere's disease, epilepsy, claustrophobia, currently pregnant or breastfeeding or planning to conceive or breastfeed during the study, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, cochlear implants, non-MR-compatible implants or devices.

xii. A history of neurological disease or injury, including a history of seizures or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion).

xiii. Unable or unwilling to fill in online questionnaires or to be contacted over the phone by study staff for periodic assessments.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
brain activation in regions of interest | baseline and 8 weeks
  Brain activation will be measured with functional magnetic resonance imaging (fMRI) during two different tasks: an interoceptive attention task and a rumination task.

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Desbordes, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States